CLINICAL TRIAL: NCT01069861
Title: A Single Arm Single Centre Study To Investigate Safety And Efficacy Of Sildenafil In Near Term And Term Newborns With Persistent Pulmonary Hypertension Of The Newborn (PPHN)
Brief Title: Study To Investigate Safety And Efficacy Of Sildenafil In The Newborns With Persistent Pulmonary Hypertension (PPHN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481276
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: PPHN; Persistent Pulmonary Hypertension of the Newborn; Hypoxic Respiratory Failure
Keywords: PPHN; neonates; sildanefil IV
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one (Experimental)
  Interventions: Drug: sildanefil

INTERVENTIONS:
Drug: sildanefil — Intravenous sildenafil citrate will be administered as a loading dose of 0.1 mg/kg given over 30 minutes. This will be followed by a maintenance treatment consisting of an intravenous infusion of 0.03 mg/kg/hr. The duration of the infusion will be determined by the need of the individual patient, but will be reviewed at Day 7 if still ongoing, and will not continue past Day 14.

SUMMARY:
Sildenafil is efficacious in newborns with persistent pulmonary hypertension and its use will reduce the need for inhaled nitric oxide.

DETAILED DESCRIPTION:
Letter to investigator dated 18 June 2012 that study was to be terminated. Study terminated due to evolved and widespread use of standard of care, relevance of study questioned. No safety reasons or issues.

ELIGIBILITY:
Inclusion Criteria:

* 72 hours of age; and > or = to 34 weeks gestational age.
* Persistent Pulmonary Hypertension of the Newborn or Hypoxic respiratory failure associated with:

  1. Idiopathic PPHN or
  2. Meconium aspiration syndrome or
  3. Sepsis or
  4. Pneumonia
* Oxygenation Index (OI) >15 and <60 calculated

Exclusion Criteria:

* Patients already receiving inhaled nitric oxide (iNO) on referral.
* Prior or immediate need for full Cardio Pulmonary Resuscitation or Extracorporeal Membrane Oxygenation (ECMO).
* Life threatening or lethal congenital anomaly.
* Large left to right intracardiac or ductal shunting (diagnosed from echocardiogram on admission to GOSH).
* Clinically significant active seizures as per clinical judgment.
* Bleeding diathesis as per clinical judgment

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Great Ormond Street Hospital, Paediatric Intensive Care, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481276&StudyName=Study%20To%20Investigate%20Safety%20And%20Efficacy%20Of%20Sildenafil%20In%20The%20Newborns%20With%20Persistent%20Pulmonary%20Hypertension%20%28PPHN%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Sildenafil citrate administered intravenously at a loading dose of 0.1 milligram per kilogram (mg/kg) over 30 minutes infusion followed by a maintenance dose of 0.03 mg/kg per hour (mg/kg/hr) intravenous infusion up to 14 days, based on the need of individual participant.
Period: Overall Study
Arm/Group | Sildenafil
Started | 4
Completed | 1
Not Completed | 3
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Did not meet entrance criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: Sildenafil citrate administered intravenously at a loading dose of 0.1 mg/kg over 30 minutes infusion followed by a maintenance dose of 0.03 mg/kg/hr intravenous infusion up to 14 days, based on the need of individual participant.
Arm/Group | Sildenafil
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: days] | 1.5 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Requiring Inhaled Nitric Oxide (iNO) or Extracorporeal Membrane Oxygenation (ECMO)
Description: Percentage of participants who required standard therapy (iNO or ECMO) after failure of study treatment.
Time Frame: From start of infusion (baseline) up to Day 14
Population: Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis due to early study termination.
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) Based on Severity
Description: AE:any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. SAE:AE resulting in any of following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience; persistent/significant disability/incapacity; congenital anomaly. Severity criteria: "mild=does not interfere with participant's usual function; moderate=interferes to some extent with participant's usual function and severe=interferes significantly with participant's usual function".
Time Frame: Baseline up to 28 days after last dose
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Abnormal Laboratory Data
Description: Criteria for potentially clinically significant (PCS) laboratory values: hematocrit 29.2 percent (%); white blood cell (WBC) count 5.0*10^3, lymphocyte absolute 0.88*10^3, total neutrophils absolute 12.07*10^3, eosinophils absolute 0.50*10^3 per cubic millimeter (/mm^3); calcium 6.8 milligram/deciliter (mg/dL); venous bicarbonate 47.0 milliequivalent/liter (meq/L).
Time Frame: Screening, once daily for 3 days, every 48 hours thereafter till the end of infusion (up to Day 14)
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Oxygenation Index at Hour 6 and 12
Description: Oxygenation Index (OI) was calculated as the product of fraction of inspired oxygen (FiO2) and Mean Airway Pressure divided by partial pressure of oxygen in arterial blood [(FiO2*Mean Airway Pressure)/PaO2] measured in centimeter of water/millimeter of mercury (cmH2O/mmHg). FiO2 is the measure of oxygen concentration that is breathed. Mean airway pressure is defined as an average of the airway pressure throughout the respiratory cycle. PaO2 is the measure of oxygen level in the arterial blood.
Time Frame: Baseline, Hour 6, 12
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Differential Saturation (Pre- And Post-ductal) at Hour 6 and 12
Description: Differential oxygenation saturation between preductal and postductal sites as measured by pulse oximetry. A difference of greater than (>) 5 percent (%) to 10% in saturation indicates right-to-left shunt through the ductus arteriosus. Oxygenation saturation is measured as percentage of hemoglobin binding sites occupied by oxygen in the blood.
Time Frame: Baseline, Hour 6, 12
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Ratio of Partial Pressure of Oxygen in Arterial Blood to the Fraction of Inspired Oxygen (P/F) at Hour 6 and 12
Description: The ratio of partial pressure of arterial oxygen and fraction of inspired oxygen is a comparison between the oxygen level in the arterial blood and the oxygen concentration that is breathed. It helps to determine the degree of any problems with how the lungs transfer oxygen to the blood.
Time Frame: Baseline, Hour 6, 12
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Mechanical Ventilation
Description: The number of days from the start to the stop of mechanical ventilation, if multiple ventilations occurred during the follow-up, the sum of the duration of each ventilation was used for analyses. Mechanical ventilation was defined as use of mechanical assistance or replacement of spontaneous breathing.
Time Frame: Baseline up to 28 days after last dose
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to Receipt of Standard Therapy (Inhaled Nitric Oxide [iNO] or Extracorporeal Membrane Oxygenation [ECMO])
Description: Time from start of treatment up to introduction of standard therapy. If participants did not receive standard therapy within 14 days after initiation of the study treatment, then Day 14 was the censoring time.
Time Frame: Baseline up to 28 days after last dose
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

9. Secondary Outcome: Population Pharmacokinetics of Sildenafil
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose, 5 and 30 minutes post-loading infusion, within 48 to 72, 96 to 120 hours during infusion, within 4 to 8, 18 to 24 and 44 to 48 hours post-maintenance infusion
Reporting Status: Not Posted

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sildenafil Metabolite (UK-103320)
Time Frame: as for outcome 9
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Duration of Study Medication
Description: The duration of the infusion was determined as per investigator's discretion up to Day 7 or Day 14.
Time Frame: Baseline up to Day 14
Population: as for outcome 1
Arm/Group | Sildenafil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sildenafil
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=4)
Congenital pneumonia (Congenital, familial and genetic disorders) | 1
Persistent foetal circulation (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=4)
Cardiac disorder (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Infusion site erythema (General disorders) | 1
Incorrect drug administration duration (Injury, poisoning and procedural complications) | 1
Blood lactic acid increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued, therefore not all data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.